CLINICAL TRIAL: NCT03591159
Title: The Effect of Membrane Sweeping on the Delivery Time and the Need of Induction in Term Pregnancy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Batuhan Turgay, MD. Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-604-18
Record Dates: First submitted 2018-06-19; First posted 2018-07-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Delivery, Obstetric

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Membrane Sweeping Group (Active Comparator)
  Interventions: Other: Membran Sweeping
- Control Group (No Intervention)

INTERVENTIONS:
Other: Membran Sweeping — Cervical Membrane Sweeping by digital examination
  Arms: Membrane Sweeping Group

SUMMARY:
Pregnancies that extend beyond 42 weeks of gestation are at an increased risk for poor fetal and maternal outcomes. For decreasing the number of these cases, some labor induction techniques are used. The status of the cervix is an indicator for the success of the induction. In these study, investigators investigate the effect of membrane sweeping on the need of induction and the delivery time in term pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Vertex presentation
* No contraindication for vaginal delivery
* No contraindication for labor induction

Exclusion Criteria:

* Active vaginal infection
* Previous uterine surgery
* Systemic disease
* Multiple pregnancy
* Fetal anomaly and suspicious fetal health status

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 256 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Need of Labor Induction. | During pregnancy. 40 weeks and 6 days for gestational age
  Patient need induction for delivery or not. If the patient reach 40 weeks 6 days for gestational age and spontaneous delivery doesn't begin spontaneously, labor induction is needed.
Duration of delivery | During delivery
  The time of the latent and active stage of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University School of Medicine Department of Obstetrics and Gynecology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At the end of the study, participant data access is possible by online.